CLINICAL TRIAL: NCT03317145
Title: Intermittent Pneumatic Compression (IPC) of the Foot Versus Geko™ Neuromuscular Electrostimulation (NMES): Comparison of Lower Limb Circulation Following Elective Total Hip Replacement (THR)
Brief Title: Lower Limb Blood Flow Geko vs Foot Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Collaborators: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FSK-FP-001
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2017-10

CONDITIONS: Venous Thrombosis; Arthroplasty, Replacement, Hip
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary embolism; neuromuscular electrostimulation; foot compression; hip replacement
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients who have had a total hip replacement will be randomised to wear either a foot compression (IPC) device or a neuromuscular electrostimulation (NMES) device (gekoTM) first. Blood flow will be measured using both devices on the same patient in sequence. The blood flow measurements will be done by ultrasound. Each ultrasound assessment will take approximately 30 minutes in total. Baseline blood flow measurements will be taken initially. The first device will then be fitted and allowed to operate for 10 minutes before ultrasound measurements are taken. After a rest period of 30 minutes, the second device is then fitted and allowed to operate for 10 minutes, following which blood flow measurements are repeated. Patients will then be asked to complete a questionnaire to assess the comfort of each device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (NMES followed by IPC) (Active Comparator): Arm A (NMES followed by IPC). Following baseline blood flow measurements using ultrasound, the neuromuscular electrostimulation (NMES) device will be fitted and allowed to operate for 10 minutes. Blood flow measurements will then be repeated. The NMES device will be removed. After a 30 minute rest period, the intermittent pneumatic compression (IPC) device will be fitted, activated for 10 minutes and then blood flow measurements repeated.
  Interventions: Device: Neuromuscular electrostimulation (NMES) device; Device: Intermittent pneumatic compression (IPC) device
- Arm B (IPC followed by NMES) (Active Comparator): Arm B (IPC followed by NMES). Following baseline blood flow measurements using ultrasound, the intermittent pneumatic compression device (IPC) will be fitted and allowed to operate for 10 minutes. Blood flow measurements will then be repeated. The IPC device will be removed. After a 30 minute rest period, the neuromuscular electrostimulation (NMES) device will then be fitted, activated for 10 minutes and then blood flow measurements repeated
  Interventions: Device: Neuromuscular electrostimulation (NMES) device; Device: Intermittent pneumatic compression (IPC) device

INTERVENTIONS:
Device: Neuromuscular electrostimulation (NMES) device — A mobile peroneal nerve stimulator
  Other Names: Geko T-1
Device: Intermittent pneumatic compression (IPC) device — A foot pump or foot compression device
  Other Names: Vadoplex

SUMMARY:
The aim of this pilot study was to assess venous flow parameters in patients following total hip arthroplasty, comparing an intermittent pneumatic compression foot device with a portable neuromuscular electrostimulator device. Assessments were performed in a single sitting before hospital discharge, between days 1 to 4 post operatively. The total duration of participation for each patient who completed the study was approximately 2.5 hours.

DETAILED DESCRIPTION:
Ethical approval was obtained from the National Research Ethics Service (Edgbaston), reference 13/WM/0139. Upon admission to hospital for THA, eligible patients were invited to participate in the study. Inclusion criteria were: patients undergoing primary THA, in good general health and fitness, age 18 years or over and the ability to provide written informed consent. Patients were taken to the ultrasound suite within the first three days following surgery.

Baseline ultrasound Patients lay in bed, the back supported at approximately 45 degrees, legs lying horizontal with their knees extended. Duplex ultrasound was then performed on the superficial femoral vein (Acuson S2000, Siemens). Baseline bilateral venous assessments of peak velocity, mean velocity, volume flow and vessel diameter were taken in triplicate. All scans were performed by the same ultrasonographer for consistency. Gate size was adjusted to just within the vessel wall.

Randomisation Following baseline measurements, patients were fitted with either the NMES device or an IPC device, the order determined by randomisation using online software. A representative from the study sponsor provided sealed envelopes containing the arm to be randomised which was opened on the day of testing.

Patients were randomised into arm A (NMES first, IPC second) or arm B (IPC first, NMES second). Blinding was not possible because the obvious physical differences between the two devices. Following testing of the first device, a 30-minute rest period was then given. The second device was then tested. All devices were fitted by the first author. All patients underwent scanning by the same sonographer to ensure consistency in data recording.

NMES application The NMES device (Geko T-1, Firstkind Ltd., High Wycombe, United Kingdom) was applied to both legs as per the manufacturer's instructions. The skin over the fibula head was prepared with an exfoliation pad, followed by an alcohol wipe. The device was applied to the skin using an adhesive strip and positioned so that the built-in electrodes were positioned over the common peroneal nerve. An overlay strip was then used to improve skin contact. A charge balanced short single pulse with a current of 27mA was delivered at a frequency of once per second. The pulse width adjustment has seven selectable stimulation settings ranging from 70 - 560 μs and was increased until a visible foot twitch was produced. Following successful application of the device for ten minutes, venous blood flow measurements were repeated.

IPC application

An IPC device (Vadoplex, OPED UK, UK) was fitted to each foot as per the manufacturer's instructions and activated for ten minutes prior to recording venous flow. The IPC provides a pump inflation pressure of 120mmHg, inflating once every 20 seconds. Each inflation was maintained for approximately 1 second, before deflation occurred. The maximum recording duration of the ultrasound scanner was 14 seconds. In order to capture 20 seconds of data, two contiguous measurements of 14 and 6 seconds were made. The machine records flow within the vessel. Since flow varies within the vessel, the machine is able to use a complex algorithm to sample velocities and flow over time and hence calculate the mean. In order to calculate mean velocity and volume flow over a complete 20 second cycle, we used the following equation:

1. Measure the blood flow during inflation (F1) and record the time duration of this flow (A).
2. Measure the blood flow during the opposite, deflated, part of the cycle (F2) and record the total cycle duration (B).

The calculation below provides a summated value for flow.

Total flow = [(A/B) x F1)] + [(1-(A/B)) x F2]

Device acceptability Patients were asked to rate comfort of the devices using a verbal rating score: 1 extremely comfortable, 2 comfortable, 3 uncomfortable, 4 very uncomfortable, 5 extremely uncomfortable.

Power analysis and statistical analysis Data from an unpublished study in healthy volunteers of the NMES device verses IPC comparing venous flow parameters, showed a significant benefit of NMES, with an effect size of 1.4 (Cohen's d). Sample size calculation based on this effect size gave a power in excess of 90% for a design of ten subjects per site.

We checked for significant association (p<0.05) of device, measurement order and leg on blood flow parameters of interest using generalized linear latent and mixed model with a random effects term to account for repeated measures on a given subject using Stata10 (Stata Corp, college station, TX). Blood flow parameters are reported as mean and 95% confidence intervals (CI). A Wilcoxon signed rank test was used to analyse the verbal rating scores for patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary THA,
* in good general health and fitness,
* age 18 years or over
* able to provide written informed consent.

Exclusion Criteria:

* Are requiring hip revision surgery
* Previous or current diagnosis of deep vein thrombosis (DVT) or pulmonary embolism (PE).
* History or signs of significant haematological disorders (especially in relation to clotting or coagulation) or thrombophlebitis.
* Peripheral arterial disease, clinically significant varicose veins or lower limb ulceration or ischemia.
* Recent surgery within the last 3 months (such as abdominal, gynaecological, hip or knee replacement).
* Recent trauma to lower limb.
* Chronic Obesity (BMI Index >40kg/m2).
* Pregnancy.
* Significant history of following diseases i. Cardiovascular: Recent MI (< 6 months) ii. Percutaneous Coronary Intervention (PCI) with stent (< 3 months for Bare metal stent (BMS) and < 12 months for Drug Eluding Stent (DES) iii. Moderate to severe CCF, uncontrolled AF iv. Neurological: Stroke, Hemiplegia/Paraplegia, Myopathies v. Renal: Moderate to severely impaired renal function vi. Hepatic: Moderate to severely impaired hepatic function vii. Psychiatric disorders viii. Dermatological conditions affecting lower limbs
* On LMWH/Heparin (Prophylactic/therapeutic doses) or Warfarin or warfarin stopped recently and replaced by LMWH/ Heparin
* Long term steroid use with dermatological changes
* A pulse rate of less than 40 beats/minute
* A sitting systolic blood pressure >180 and <100 mmHg and/or a sitting diastolic pressure of >100 mmHg.
* Participation in any clinical study during the eight (8) weeks preceding the screening period
* THR done for hip fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-24 (Actual); Primary Completion 2014-02-19 (Actual); Study Completion 2014-02-19 (Actual)

PRIMARY OUTCOMES:
Venous flow at baseline | "t0" - 30 minutes to include the ultrasound assessment, performed between days 1 and 4 post operatively
  Measured within the superficial femoral vein using ultrasound
Venous flow after application of device 1 | "t1" - 90 minutes to include the ultrasound assessment
  Measured within the superficial femoral vein using ultrasound
Venous flow after application of device 2 | "t2" - 150 minutes to include the ultrasound assessment
  Measured within the superficial femoral vein using ultrasound

SECONDARY OUTCOMES:
Patient satisfaction with device 1 | Immediately after completion of the ultrasound assessment for device 1, at "t1" - 90 minutes
  verbal rating score: 1 extremely comfortable, 2 comfortable, 3 uncomfortable, 4 very uncomfortable, 5 extremely uncomfortable.
Patient satisfaction with device 2 | Immediately after completion of the ultrasound assessment for device 2, at "t2" - 150 minutes
  verbal rating score: 1 extremely comfortable, 2 comfortable, 3 uncomfortable, 4 very uncomfortable, 5 extremely uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Stranks, FRCS, Principal Investigator — North Hampshire Hospital, Basingstoke

IPD SHARING:
Plan to Share IPD: No
We would be happy to share individual participant data if requested by other researchers although have no formal plans to publish this at present. All data shared would be anonymised.

REFERENCES:
- [Background] Warwick DJ, Shaikh A, Gadola S, Stokes M, Worsley P, Bain D, Tucker AT, Gadola SD. Neuromuscular electrostimulation viathe common peroneal nerve promotes lower limb blood flow in a below-kneecast: A potential for thromboprophylaxis. Bone Joint Res. 2013 Sep 2;2(9):179-85. doi: 10.1302/2046-3758.29.2000176. Print 2013. PMID 23999610
- [Background] Williams KJ, Moore HM, Davies AH. Haemodynamic changes with the use of neuromuscular electrical stimulation compared to intermittent pneumatic compression. Phlebology. 2015 Jun;30(5):365-72. doi: 10.1177/0268355514531255. Epub 2014 Apr 10. PMID 24722790